CLINICAL TRIAL: NCT07006896
Title: Labor Induction After Cesarean: A Randomized Trial Of Cervical Balloon With or Without Oxytocin
Brief Title: Induction of Labor After Cesarean Using Foley Alone vs. Concurrent Foley and Oxytocin
Acronym: LIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Lisa Levine, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 858270
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Labor Induction; Cesarean Delivery
Keywords: Labor; Induction; Cesarean; TOLAC; Foley; Oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent Foley balloon and Oxytocin (Experimental): Cervical ripening will begin with a Foley balloon and concurrent oxytocin, started within 2 hour of balloon placement
  Interventions: Device: Foley balloon; Drug: Oxytocin
- Foley balloon alone (Active Comparator): Cervical ripening will begin with a Foley balloon alone. Oxytocin will not be started until the balloon is removed or expelled, though can be considered if the balloon remains in place for >8 hours
  Interventions: Device: Foley balloon

INTERVENTIONS:
Device: Foley balloon — Foley balloon for induction of labor
  Other Names: Foley catheter; Cervical ripening balloon
Drug: Oxytocin — Pitocin for induction of labor
  Other Names: Pitocin
  Arms: Concurrent Foley balloon and Oxytocin

SUMMARY:
A randomized trial of patients undergoing a term (≥37 weeks) induction of labor with a history of one prior Cesarean delivery, wherein the provider intends to use a Foley catheter for cervical ripening. The investigators will be comparing Foley alone with concurrent Foley and Oxytocin use at the start of the induction. With this trial, the investigators aim to test our central hypothesis that concurrent Foley and Oxytocin will decrease time to delivery without increasing risks, compared to Foley alone.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for induction of labor
* Live singleton gestation ≥37 weeks
* History of 1 cesarean delivery
* ≥18 years of age
* Cephalic presentation
* Intact membranes
* English or Spanish speaking (Able to read/understand consent and instructions)
* Cervical dilation <3cm and Bishop score <8

Exclusion Criteria:

* >1 prior Cesarean delivery
* Known chorioamnionitis
* Major fetal anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Time to delivery | At delivery
  The primary endpoint will be time from start of induction until delivery (hours)

SECONDARY OUTCOMES:
Estimated postpartum blood loss | At delivery
  Estimated postpartum blood loss in mL
Postpartum hemorrhage | Within 6 weeks of delivery
  Estimated blood loss≥ 1L
Number of Participants with Chorioamnionitis | At delivery
  Documented chorioamnionitis
Mode of delivery | At delivery
  Successful vaginal birth after cesarean (VBAC) or repeat cesarean delivery (rCD)
Number of Participants with Uterine Rupture | At delivery
  Uterine rupture noted at the time of cesarean delivery
Maternal morbidity | Within 6 weeks of delivery
  Defined as a composite endpoint consisting of at least one occurrence of the following outcomes: postpartum hemorrhage, blood transfusion, endometritis, wound/laceration breakdown or infection, venous thromboembolism and hospital readmission with 6 weeks
Neonatal morbidity | Within 6 weeks of delivery
  Defined as neonatal resuscitation requiring supplemental oxygen outside of the delivery room for at least 12 hours of culture proven/presumed neonatal sepsis
Maternal length of stay | From date of delivery to date of discharge from hospital postpartum, up to 6 weeks from delivery
  Measured by hours from admission to postpartum discharge
Neonatal length of stay | From date of delivery to date of discharge from hospital postpartum, up to 6 weeks from delivery
  Length of stay from birth to discharge, measured in hours
NICU stay greater than 48 hours | From date of delivery to date of discharge from hospital postpartum, up to 6 weeks from delivery
  Admission to the NICU for more than 48 hours
Maternal patient satisfaction as measured by the Hollins Martin Birth Satisfaction scale-Revised (BSS-R) | From time of delivery to discharge from hospital, up to 6 weeks from delivery
  Patient satisfaction as measured by the BSS-R with a possible score of 0-40 with 0 equaling the least birth satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Levine, MD MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Hollis S, Campbell F. What is meant by intention to treat analysis? Survey of published randomised controlled trials. BMJ. 1999 Sep 11;319(7211):670-4. doi: 10.1136/bmj.319.7211.670. PMID 10480822
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Levine LD, Downes KL, Hamm RF, Srinivas SK. Evaluating the impact of a standardized induction protocol to reduce adverse perinatal outcomes: a prospective cohort study. J Matern Fetal Neonatal Med. 2021 Oct;34(19):3200-3207. doi: 10.1080/14767058.2019.1680629. Epub 2019 Oct 24. PMID 31645154
- [Background] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571
- [Background] Jamaluddin A, Azhary JMK, Hong JGS, Hamdan M, Tan PC. Early versus delayed amniotomy with immediate oxytocin after Foley catheter cervical ripening in multiparous women with labor induction: A randomized controlled trial. Int J Gynaecol Obstet. 2023 Feb;160(2):661-669. doi: 10.1002/ijgo.14361. Epub 2022 Aug 8. PMID 35869943
- [Background] Gomez Slagle HB, Fonge YN, Caplan R, Pfeuti CK, Sciscione AC, Hoffman MK. Early vs expectant artificial rupture of membranes following Foley catheter ripening: a randomized controlled trial. Am J Obstet Gynecol. 2022 May;226(5):724.e1-724.e9. doi: 10.1016/j.ajog.2021.11.1368. Epub 2022 Feb 6. PMID 35135684
- [Background] Secchi D, Alberic J, Gobillot S, Ghenassia A, Roustit M, Chauleur C, Hoffmann P, Raia-Barjat T. Balloon catheter vs oxytocin alone for induction of labor in women with one previous cesarean section and an unfavorable cervix: a multicenter, retrospective study. Arch Gynecol Obstet. 2022 Aug;306(2):379-387. doi: 10.1007/s00404-021-06298-y. Epub 2021 Oct 28. PMID 34708257
- [Background] Hoffman MK, Hunter Grant G. Induction of labor in women with a prior cesarean delivery. Semin Perinatol. 2015 Oct;39(6):471-4. doi: 10.1053/j.semperi.2015.07.011. Epub 2015 Sep 11. PMID 26365010
- [Background] West HM, Jozwiak M, Dodd JM. Methods of term labour induction for women with a previous caesarean section. Cochrane Database Syst Rev. 2017 Jun 9;6(6):CD009792. doi: 10.1002/14651858.CD009792.pub3. PMID 28599068
- [Background] Kehl S, Weiss C, Rath W. Balloon catheters for induction of labor at term after previous cesarean section: a systematic review. Eur J Obstet Gynecol Reprod Biol. 2016 Sep;204:44-50. doi: 10.1016/j.ejogrb.2016.07.505. Epub 2016 Aug 3. PMID 27521597
- [Background] Levin G, Tsur A, Burke YZ, Meyer R. Methods of induction of labor after cesarean with no prior vaginal delivery-Perinatal outcomes. Int J Gynaecol Obstet. 2023 Feb;160(2):612-619. doi: 10.1002/ijgo.14318. Epub 2022 Jul 14. PMID 35751576
- [Background] Landon MB, Hauth JC, Leveno KJ, Spong CY, Leindecker S, Varner MW, Moawad AH, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai B, Langer O, Thorp JM, Ramin SM, Mercer BM, Gabbe SG; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Maternal and perinatal outcomes associated with a trial of labor after prior cesarean delivery. N Engl J Med. 2004 Dec 16;351(25):2581-9. doi: 10.1056/NEJMoa040405. Epub 2004 Dec 14. PMID 15598960
- [Background] Deshmukh U, Denoble AE, Son M. Trial of labor after cesarean, vaginal birth after cesarean, and the risk of uterine rupture: an expert review. Am J Obstet Gynecol. 2024 Mar;230(3S):S783-S803. doi: 10.1016/j.ajog.2022.10.030. Epub 2023 Jul 13. PMID 38462257
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Bruno AM, Allshouse AA, Metz TD. Trends in Attempted and Successful Trial of Labor After Cesarean Delivery in the United States From 2010 to 2020. Obstet Gynecol. 2023 Jan 1;141(1):173-175. doi: 10.1097/AOG.0000000000004998. Epub 2022 Nov 30. PMID 36701618
- [Background] ACOG Practice Bulletin No. 205: Vaginal Birth After Cesarean Delivery. Obstet Gynecol. 2019 Feb;133(2):e110-e127. doi: 10.1097/AOG.0000000000003078. PMID 30681543
- [Background] Stephenson J. Rate of First-time Cesarean Deliveries on the Rise in the US. JAMA Health Forum. 2022 Jul 1;3(7):e222824. doi: 10.1001/jamahealthforum.2022.2824. No abstract available. PMID 36219002